CLINICAL TRIAL: NCT01343992
Title: Evaluation of the Influence of Bed Rest After Embryo Transfer in Outcome of IVF Treatment With Ovum Donation.
Brief Title: Bed Rest or no Bed Rest?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Jose Remohi, Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0912-C-065-SA
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: In Vitro Fertilization
Keywords: Embryo transfer; Implantation rate; Pregnancy rate; bedrest; neutral; benevolent; deterious; implantation; gestation rates
MeSH Terms: interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bedrest (Active Comparator): Patients will rest in bed ten minutes after the embryo transfer.
  Interventions: Behavioral: Bed rest
- No bed rest (Experimental): Patients will not rest after the embryo transfer.
  Interventions: Behavioral: No bedrest

INTERVENTIONS:
Behavioral: Bed rest — Patients will rest in bed ten minutes after the embryo transfer.
  Arms: Bedrest
Behavioral: No bedrest — Patients will not rest in bed after the embryo transfer.
  Arms: No bed rest

SUMMARY:
A comparative study to determine whether bed rest after embryo transfer (ET) affects on IVF (In Vitro Fertilization)outcome. This study includes 240 patients undergoing IVF treatment with donated oocytes. All the procedures of IVF, of the embryo transfer, and of the administration of medications are performed as always and there are no variations. The only highlighted procedure in this study is immediately after the embryo transfer. There are two groups: one which will rest in bed for 10 minutes after the transfer and one which will not rest after the transfer. Both procedures are common, usually depending on the habitual clinical practice of each clinic internationally. Patients from both group receive the routine post transfer instructions and treatment.

ELIGIBILITY:
Inclusion criteria:

* Infertile Patients with fertility problems due to tubaric or ovarian problems with normozoospermatic couple
* Patient and her couple with ages between ages 20 - 49 years old
* BMI < 25 kg/m2
* IVF treatment with oocyte donation
* Elective transfer of 2 embryos of day 3 embryos or day 5/6 embryos transferred
* First cycle of embryo transfer

Exclusion criteria:

* Patients with uterine abnormalities, significant uterine fibroids, Hydrosalphinx
* History of recurrent pregnancy loss
* severe male factor were excluded from the study

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Live birth infant rate after delivery from both groups of study | 10 months
  Whether bed rest after embryo transfer affects the pregnancy rate in IVF treatment with oocyte donation.

SECONDARY OUTCOMES:
Implantation rate | 2 months
Miscarriage rate | 5 months
Birth weight of live newborn infant after delivery | 10 months
Birth height of live newborn infant after delivery | 10 months
Cranial perimeter of live newborn infant after delivery | 10 months
APGAR score of live newborn infant after delivery | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sharayi Gaikwad, MD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Spain

REFERENCES:
- [Derived] Gaikwad S, Garrido N, Cobo A, Pellicer A, Remohi J. Bed rest after embryo transfer negatively affects in vitro fertilization: a randomized controlled clinical trial. Fertil Steril. 2013 Sep;100(3):729-35. doi: 10.1016/j.fertnstert.2013.05.011. Epub 2013 Jun 10. PMID 23755954